CLINICAL TRIAL: NCT00186030
Title: Reducing Risk and Trauma-Related Stress in Persons Living With HIV
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R03MH063643-02 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2005-09

CONDITIONS: HIV; PTSD
Keywords: HIV; AIDS; PTSD; Prevention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Acquired Immunodeficiency Syndrome

INTERVENTIONS:
Behavioral: HIV Skills-based Prevention

SUMMARY:
This two-year study tested the concept that an intervention, which reduces trauma-related symptoms among adults who are living with human immunodeficiency virus (HIV), are experiencing trauma-related stress symptoms, and engaging in behavior that facilitates HIV transmission, can reduce the transmission risk of (HIV). Our central premise was that by first treating trauma symptoms, we would enhance the effects of a skills-building HIV risk reduction intervention for adults experiencing trauma-related symptoms such as hyperarousal, dissociation, and avoidance.

The study aims were to:

1. To determine if decreasing trauma-related stress symptoms improves HIV risk reduction behavior above a standard HIV risk reduction intervention alone post-intervention and 3 months after the small group intervention sessions;
2. To determine whether key variables moderate the intervention's effects. For instance, gender, age, ethnicity, or psychological distress (e.g., depression, anxiety) may interact with the intervention to affect risky sexual or drug-related behavior; and
3. To determine whether there is evidence that the theoretical mediator variables, which include trauma-related stress symptoms, self-efficacy, communication skills, and social support mediate the intervention's effects on outcomes. This information addresses the theoretical question of why the intervention works.

DETAILED DESCRIPTION:
There are no published longitudinal studies examining the impact of traumatic events on risk behavior among HIV-positive men and women. As a result, we know very little about how stress, particularly trauma-related stress, influences HIV risk behavior. This study will be one of the first randomized studies to examine the efficacy of reducing HIV risk behavior by combining a trauma-focused stress reduction intervention with a standard HIV prevention skills intervention. This study is specifically targeting a low-income, urban population, a group that experiences a disproportionate rate of crime as well as HIV infection. Findings of the research will likely provide information on the relationship between trauma and risk behavior. Furthermore, this research can identify key issues related to stress, psychosocial factors, and overall health that will be relevant to investigate in future, larger-scale studies of HIV-positive as well as HIV-negative populations.

Individuals who reported living with HIV, engaging in HIV risk behavior in the past 3 months, experiencing a traumatic stressor and trauma-related symptoms in the past 3 months were assigned to one of three conditions: 1) standard HIV prevention skills; 2) standard HIV prevention skills + trauma-focused stress reduction skills training; or 3) trauma-focused stress reduction skills training.

ELIGIBILITY:
Inclusion Criteria:

* must be 18 years or older, must be HIV-positive
* report engaging in behavior that could put them at risk for HIV transmission during the past 3 months
* report experiencing one or more trauma-related symptoms (i.e., reexperiencing, hyperarousal, or avoidance) occurring within the past three months.

Exclusion Criteria:

* experience psychological symptoms or substance use problems so severe that it would impair their ability or the ability of others to participate in a group intervention

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2003-04; Study Completion 2004-03

PRIMARY OUTCOMES:
To determine if decreasing trauma-related stress symptoms improves HIV risk reduction behavior above a standard HIV risk reduction intervention alone post-intervention and 3 months after the small group intervention sessions

SECONDARY OUTCOMES:
To determine whether key variables moderate the intervention's effects. For instance, gender, age, ethnicity, or psychological distress (e.g., depression, anxiety) may interact with the intervention to affect risky sexual or drug-related behavior.
To determine whether there is evidence that the theoretical mediator variables, which include trauma-related stress symptoms, self-efficacy, communication skills, and social support mediate the intervention's effects on outcomes. This information will

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Gore-Felton, PhD, Principal Investigator — Stanford University
Locations (1):
- Center for AIDS Intervention Research (CAIR), Milwaukee, Wisconsin, United States